CLINICAL TRIAL: NCT03043170
Title: Diagnostic Investigation and Prediction of Shock (The DiPS Study)
Brief Title: Diagnostic Investigation and Prediction of Shock
Acronym: DiPS
Status: Completed | Type: Observational
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: CardiffU
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Shock
Keywords: Adults; Emergency Department; Haemodynamics; Resuscitation; Shock; Uscom
MeSH Terms: conditions — Shock; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound Cardiac Output Monitor — a device for assessing haemodynamics continuously and non-invasively using Doppler wave ultrasound
  Other Names: USCOM®; USCOM Pty Ltd, NSW, Australia

SUMMARY:
Background to the research Patients present to Emergency Departments (ED) with a spectrum of illness, many of which are life- threatening. The body has the ability to compensate in the early stages when things go wrong so that on the surface patients do not appear as sick as they really are. Under-diagnosis of severity of illness leads to under-treatment, unnecessary mortality, and unnecessary hospital costs. Earlier diagnosis and consequent treatment will result in prudent healthcare, cost-benefit and better patient outcomes.

Evaluating the true underlying patient haemodynamics such as cardiac output, cardiac power and peripheral pressures gives vital clues to the hidden seriousness of illness and is a guide to better management. Few EDs in the world assess such haemodynamics. After evaluating a haemodynamic protocol one centre in Australia was able to reduce its death rate for septic shock at 30 days from 38% to 7%. We would like to evaluate whether the same would occur if applied across EDs in Wales. However, before we can do that we need to strengthen our understanding of haemodynamics, and of relevant protocols and non-invasive devices that help us to acquire such information.

Study Design After ethics and institutional approval is obtained from we will conduct a prospective, single-centre, cohort study on 354 adult patients with possible shock associated with an acute illness or injury who present to the Emergency Department of the University Hospital of Wales, and follow them up for 7 days. 354 is a credible number to confirm that the strategy works.

Written consent will be obtained either from the patient or a relative wherever possible but a waiver of consent apply to patients who, because of confusion, unconsciousness or severe disability, may be unable to give consent. In these cases, consent will first be sought from a second doctor and/or nurse. Thereafter, consent will be obtained from the patient or a relative as soon as practically possible.

What you hope to discover

We expect to discover that:

* Uscom variables predict 7-day survival and ICU admission
* Uscom variables improve the detection and classification of shock
* The LiPS definition can be improved.
* The objective definition is better than doctors experience
* Patients have a good experience and are satisfied with care

DETAILED DESCRIPTION:
Patients frequently present to emergency departments (EDs) with critical illness and injury. Shock is a life-threatening emergency, which requires urgent and rapid assessment, diagnosis and treatment, and can be classified into distributive-septic (62%), distributive-non-septic (4%), hypovolaemic (16%), cardiogenic (16%) and obstructive (2%). Sepsis is the leading cause of in-hospital death, and approximately 80% of these patients are admitted through the ED. In Chinese patients presenting to an ED in Hong Kong we have previously derived and validated a simple, a priori, pragmatic, quantitative method for recognising and classifying shock - Li's Practical Shock (LiPS) tool. This method has been validated against ICU admission and early mortality. However, it was derived in a single population in a single centre, and requires further validation and refined in other settings. Further, it does not sub-classify patients beyond 'normal, cold and warm shock', does not guide next steps in treatment, and the assessment of the peripheries is very subjective.

Evaluating the true underlying patient haemodynamics such as cardiac output, cardiac power and peripheral pressures gives vital clues to the hidden seriousness of illness and is a guide to better management. Few EDs in the world assess such haemodynamics. After evaluating a haemodynamic protocol one centre in Australia was able to reduce its death rate for septic shock at 30 days from 38% to 7%. We would like to evaluate whether the same would occur if applied across EDs in Wales. However, before we can do that we need to strengthen our understanding of haemodynamics, and of relevant protocols and non-invasive devices that help us to acquire such information.

There are many unanswered questions such as:

* Do Uscom-derived haemodynamic variables measured in the ED predict patients who at high risk of death, admission to ICU, and have shock?
* Does a refined LiPS definition better predict mortality and ICU admission?
* Do advanced haemodynamic predictors and/or refined LiPS predict better than experienced physicians the presence and classification of patients with shock, mortality and ICU admission?

This study will answer two main questions:

1. What is the probability that a patient has shock?
2. What type of shock does the patient have?

We propose:

1. To investigate whether advanced haemodynamic variables using USCOM predict 7-day mortality and ICU admission.
2. To investigate whether advanced haemodynamic variables using USCOM improve the detection and classification of shock.
3. To validate and refine Li's a priori Pragmatic Shock (LiPS) method for detecting and classifying shock.
4. To evaluate clinical experience for shock.
5. To inform on the feasibility of future studies

After ethics and institutional approval is obtained from we will conduct a prospective, single-centre, cohort study on 354 adult patients with possible shock associated with an acute illness or injury who present to the Emergency Department of the University Hospital of Wales, and follow them up for 7 days. 354 is a credible number to confirm that the strategy works.

Written consent will be obtained either from the patient or a relative wherever possible but a waiver of consent apply to patients who, because of confusion, unconsciousness or severe disability, may be unable to give consent. In these cases, consent will first be sought from a second doctor and/or nurse. Thereafter, consent will be obtained from the patient or a relative as soon as practically possible.

The challenge is to discover a strategy that has a sensitivity >67% and specificity >72% for determining in-hospital mortality in clinically deteriorating or potentially shocked patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years
* a NEWS≥3,
* requiring a trolley

Exclusion Criteria:

• <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients presenting to the ED of University Hospital of Wales (UHW) with a NEWS>3, requiring a trolley, and during research study periods
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Composite of ICCU/all cause mortality | 7 days
  Number of patients with admission to either ICU, or CCU, or death from any cause

SECONDARY OUTCOMES:
In-hospital mortality | 28 days
  Number of patients with death from any cause in hospital
28-day mortality | 28 days
  Number of patients with death from any cause within 28 days
Admission to ICCU | 7 days
  Number of patients with admission to either ICU or CCU
ED shock | Within 4 hours of ED arrival
  Number of patients with shock in the ED defined according to LiPS criteria
Types of ED Shock | Within 4 hours of ED arrival
  Number of patients with ED shock categorised as either primarily restrictive or hypovolaemic, or cardiogenic or obstructive shock.

OTHER OUTCOMES:
Feasibility variables | 4 hours
  patient acceptance and experience, medical and nursing acceptance and experience, and evaluation of the infrastructure necessary to perform future definitive randomised controlled trials of this type in the emergency setting, to inform on sample sizes for future studies, to assess the processes and workload involved in patient recruitment, consent and reasons for non-participation, and to assess the potential loss to follow up and impact on analysis and interpretation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Rainer, MD, Principal Investigator — Professor of Emergency Medicine
Locations (1):
- Cardiff University, Cardiff, S Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No plan